CLINICAL TRIAL: NCT04070781
Title: Phase I Study of Itacitinib in Combination With Tocilizumab for the Treatment of Steroid Refractory Acute Graft Versus Host Disease
Brief Title: Itacitinib and Tocilizumab for Steroid Refractory Acute Graft Versus Host Disease
Acronym: GVHD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The primary reason for study closure is slow enrollment.
Sponsor: Columbia University (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAR8757
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Steroid Refractory GVHD; Graft Vs Host Disease
Keywords: Steroid Refractory GVHD
MeSH Terms: conditions — Graft vs Host Disease | interventions — itacitinib; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Itacitinib + Tocilizumab (Experimental): A dose de-escalation design will be used to identify the MTD of both itacitinib and tocilizumab when given in combination. The following two levels will be tested with at least 6 patients per dose:
  * Dose level 1: Itacitinib 200 mg daily + tocilizumab 8mg/kg on cycle 1, day 1 (can repeat cycle 2 day 1 if Partial Response (PR) - Starting dose level
  * Dose level -1: Itacitinib 200 mg daily + tocilizumab 4mg/kg on cycle 1, day 1 (can repeat cycle 2 day 1 if Partial Response (PR) - Dose De-escalation level
  Itacitinib will be given daily in 28-day long cycles, tocilizumab will be given every 4 weeks in 28-day cycles.
  Interventions: Drug: Itacitinib; Drug: Tocilizumab
- Dose Expansion (Experimental): Once the MTD is determined, an additional 10 patients as an expansion cohort to further define the safety profile of the combination and estimate its response rate.
  Interventions: Drug: Itacitinib; Drug: Tocilizumab

INTERVENTIONS:
Drug: Itacitinib — Itacitinib is a novel, potent, and selective inhibitor of the Janus Kinase (JAK) family of protein tyrosine kinases (TYKs) with selectivity for Janus Kinase 1 (JAK1). Itacitinib is an investigational product.
  Itacitinib 200 mg daily in 28-day long cycles
  Other Names: Itacitinib adipate
Drug: Tocilizumab — Tocilizumab is a biologic medication currently approved to treat adults with moderately to severely active rheumatoid arthritis (RA), adults with giant cell arteritis (GCA), and children ages two and above with Polyarticular Juvenile Idiopathic Arthritis (PJIA) or Systemic Juvenile Idiopathic Arthritis (SJIA). Tocilizumab blocks the inflammatory protein interleukin 6 (IL-6). This improves joint pain and swelling from arthritis and other symptoms caused by inflammation.
  Tocilizumab 4 or 8mg/kg cycle 1 day 1 every 4 weeks in 28-day cycles
  Other Names: Actemra

SUMMARY:
The study's primary objective is designed to assess the safety and tolerability, and determine the maximum tolerated dose (MTD) of both itacitinib and tocilizumab when given in combination to patients with steroid-refractory acute graft versus host disease (SR-aGVHD).

The study's secondary objectives are to:

* Estimate the day 28 response rate (ORR) [complete response (CR), very good partial response (VGPR), and partial response (PR)] of the combination of itacitinib and tocilizumab for the treatment of SR-aGVHD
* Estimate the time to response and duration of response
* Estimate the incidence of primary disease relapse while on study treatment
* Estimate the incidence of infections including viral reactivation, bacterial infections and fungal infections while on study treatment
* Estimate the progression-free survival (PFS), overall survival (OS), non-relapse mortality, GVHD-related mortality of study subjects
* Estimate the proportion of patients who successfully discontinue steroids by 6 months and 12 months after therapy initiation

DETAILED DESCRIPTION:
The treatment of acute and chronic GVHD consists mostly of steroids which has changed very little over the past 40 years. Response to current therapy for GVHD is far from perfect; only about 50% of patients respond to therapy and many of those responses are not durable.

The current study is a phase I study dose de-escalation study where up to 6 patients will be enrolled into each dose level (2 levels), followed by an expansion cohort at the MTD. The goal of the study is to determine the maximum tolerated dose of the combination of itacitinib and tocilizumab. Once the MTD is determined, the investigator will enroll 10 additional patients as an expansion cohort to further define the safety profile of the combination and estimate its response rate.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women who are at least 18 years of age
* Recipients of their first allogeneic hematopoietic stem cell transplant from any donor source (including bone marrow, mobilized peripheral blood, cord blood) and human leukocyte antigen (HLA)-match (includes matched related, matched unrelated, mismatched unrelated, and haploidentical)
* Recipients of allogeneic stem cell transplant after any conditioning regimen intensity and those who have received any GVHD prophylaxis regimen, unless it included tocilizumab and/or itacitinib
* Steroid refractory acute GVHD (SR-aGVHD) that has been clinically diagnosed as per the MAGIC criteria and/or pathologically confirmed. Biopsies should be attempted whenever possible according to the investigator's discretion but it is not required as long as alternative diagnoses such as infection or medication side effects have been adequately ruled out. SR-aGVHD is defined as acute GVHD that has failed to exhibit a response after treatment for at least 7 days with a corticosteroid dose of 2 mg/kg of methylprednisolone or prednisone equivalent. SR-aGVHD is also defined as GVHD that flares when steroids are tapered prohibiting further taper.
* Adequate renal function determined by creatinine clearance ≥ 40 mL/min measured or calculated by Cockcroft-Gault equation.
* Absence of history of irreversible liver disease such as cirrhosis or veno-occlusive disease (VOD) that has not responded to therapy
* Total bilirubin and/or transaminases (AST and/or ALT) that are ≤2.5 above institutional upper limit of normal that is not attributable to acute GVHD by biopsy
* Non-pregnant females or men and women willing to avoid pregnancy or fathering a child as evidenced by negative pregnancy test (females), non-childbearing potential (history of hysterectomy, oophorectomy, amenorrhea for 12 months) or agree to use barrier or chemical contraception for the duration of the study.
* Ability to swallow oral medication
* Able to give consent and comply with study visits and procedures

Exclusion Criteria:

* Primary disease not in complete remission, requiring active treatment, or having required treatment for relapsed disease
* Uncontrolled bacterial, viral, or fungal infections which is evidenced by hemodynamic instability, new radiological findings, new signs or symptoms, or persistently positive blood cultures as determined by the investigator.
* History of viral infection with HIV
* History of infection or exposure to hepatitis B or C with a risk of infection reactivation
* History of active or latent tuberculosis infection that has not been adequately treated
* Use of any JAK inhibitor or IL-6 antagonists for therapy or prophylaxis of acute GVHD. Continuation of calcineurin inhibitors intended for GVHD prophylaxis is allowed. Resumption of therapeutic dosing of calcineurin inhibitors that is being tapered is also allowed.
* Severe organ dysfunction unrelated to GVHD that includes cholestatic disorders or unresolved VOD (defined as ongoing organ dysfunction and bilirubin elevation unrelated to GVHD > 2.5 the institutional upper limit of normal), clinically significant or uncontrolled cardiac disease (including unstable angina, acute myocardial infarction within 6 months of enrollment, New York Heart Association, Class III or IV congestive heart failure, circulatory collapse requiring vasopressor or inotropic support, or arrhythmia that requires therapy) or clinically significant respiratory disease that requires mechanical ventilation support or 50% or greater supplemental oxygen..
* Receipt of live attenuated vaccine or the need for such a vaccine during the duration of the study
* Treatment with any other investigational agent within 7 days of enrollment (or 5 half-lives, whichever is greater)
* Treatment with any JAK inhibitor or IL-6 antagonist after stem cell transplant. Treatment with a JAK inhibitor before transplant is allowed. Treatment with IL-6 antagonist before transplant is allowed only if last dose was at least 4 weeks prior to transplant.
* Known allergies or sensitivities to itacitinib or tocilizumab
* Pregnant, breast-feeding, or unwilling or unable to avoid pregnancy or fathering a child. Pregnant women are excluded from this study as animal studies have shown that tocilizumab crosses the placenta and can interfere with fetal development in animal studies. Furthermore, itacitinib has been associated with embryo-fetal toxicity in animal studies

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
MTD of Tocilizumab IV infusion when given with Itacitinib | 28 - 35 days after the End of Treatment (EOT) or the date of the last dose of the study drug
  Maximum Tolerated Dose (MTD) is the highest dose of a drug or treatment that does not cause unacceptable side effects.
Access Safety and Tolerability | End of Cycle 1 (approximately 28 days)
  The safety and tolerability of study treatment is measured by the frequency and severity of adverse events and serious adverse events.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | End of Cycle 1 (approximately 28 days)
  The percentage of patients whose cancer shrinks or disappears after treatment (combination of itacitinib and tocilizumab for the treatment of SR-aGVHD), this will include patients with complete response (CR), very good partial response (VGPR) and partial response (PR). This rate will estimated after 28 days on treatment.
Time to Response | Up to 36 months
  Time to response as defined in the May 2009 CIBMTR Acute Graft-versus-Host Disease (GVHD) Workshop as the time needed for resolution of GVHD symptoms. Response evaluation will be relative to the assessment on Day 1.
Duration of Response | Up to 36 months
  Duration of response is defined as the interval from day 28 to progression as outlined in the May 2009 Center for International Blood and Marrow Transplant Research (CIBMTR) Acute Graft-versus-Host Disease (GVHD) Workshop
Incidence of Disease Relapse | Up to 36 months
  The occurrence of the return of a disease.
Incidence of Infections | Up to 36 months
  The occurrence of infections including viral reactivation, bacterial infections and fungal infections while on study treatment
Progression-Free Survival (PFS) | Up to 36 months
  Progression-free survival (PFS) (time alive without GVHD) probabilities will be estimated using Kaplan-Meier method, and, if exists, median with 95% confidence interval (CI) will also be reported
Overall Survival (OS) | Up to 36 months
  The length of time from the start of treatment that subjects with the disease are still alive.
Proportion of Patients Discontinuing Steroids | 6-12 months
  The proportion of patients who successfully discontinue steroids by 6 months and 12 months after therapy initiation

CONTACTS AND LOCATIONS:
Overall Officials: Markus Mapara, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York

REFERENCES:
- See also: Columbia University Medical Center — https://www.cuimc.columbia.edu/